CLINICAL TRIAL: NCT02183805
Title: Phase II Study of Chemotherapy Followed by Peripheral Stem Cell Transplantation as First Line Therapy for Metastatic Triple-negative Breast Cancer
Brief Title: Chemotherapy Followed by Peripheral Stem Cell Transplantation in Treating Metastatic Triple-negative Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty accruing subjects the study accrual was closed
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-004
Record Dates: First submitted 2014-07-01; First posted 2014-07-08 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Carcinoma Breast Stage IV
Keywords: triple negative breast cancer; autologous hematopoietic stem-cell transplantation
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Albumin-Bound Paclitaxel; CAC protocol; Cyclophosphamide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metastatic triple negative breast cancer (Experimental): Abraxane,Cyclophosphamide,Carboplatin
  Interventions: Drug: Abraxane,Cyclophosphamide,Carboplatin

INTERVENTIONS:
Drug: Abraxane,Cyclophosphamide,Carboplatin — High dose chemotherapy: Abraxane, Cyclophosphamide, Carboplatin
  Other Names: Abraxane 800 mg/m2; Cyclophosphamide 3g/m2; Carboplatin 800 mg/m2

SUMMARY:
Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

DETAILED DESCRIPTION:
To explore the progression-free survival of patients with metastatic triple-negative breast cancer treated with peripheral blood stem cell transplant (PBSCT) followed by high dose chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Histologically or cytologically proven diagnosis of breast cancer with evidence of locally recurrent or metastatic disease.
* Documentation of estrogen and progestin receptor (ER/PR) negative status and HER2/neu receptor negative status (ie, FISH negative or immunohistochemistry 0 or +1).
* Obtained complete response or Good partial response after first line chemotherapy.
* Normal organ function required prior to study entry.
* Willingness to comply with treatment plans and other study procedures.

Exclusion Criteria:

* Uncontrolled central nervous system (CNS) involvement with disease
* Fertile women unwilling to use contraceptive techniques during treatment
* Females who are pregnant
* Organ dysfunction.
* Patients may not be receiving any other investigational agents.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-06-17 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Progression free Survival | 24 months

SECONDARY OUTCOMES:
Overall Survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-Yu Yuan, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No